CLINICAL TRIAL: NCT04225546
Title: Relationship Between Sit to Stand Movement, Trunk Control and Selective Motor Control of Lower Extremity in Children With Hemiplegic and Diplegic Cerebral Palsy
Brief Title: Sit to Stand Movement in Children With Cerebral Palsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2019.261
Record Dates: First submitted 2020-01-04; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy, Spastic; Cerebral Palsy, Spastic, Diplegic
Keywords: cerebral palsy; selective control; trunk; sit to stand
MeSH Terms: conditions — Cerebral Palsy; Cerebral palsy, spastic, diplegic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient group: Patients with hemiplegic and diplegic cerebral palsy between 4 - 10 years of age
- Control group: Healthy volunteer typically developing peers

SUMMARY:
The aim of this study is to examine the relationship between trunk control and lower extremity selective motor control during the movement of sit to stand (STS) in children with cerebral palsy (CP).

DETAILED DESCRIPTION:
The aim of this study is to examine the relationship between trunk control and lower extremity selective motor control and balance problems during the movement of sit to stand (STS) frequently encountered in children with cerebral palsy (CP) in daily life and to compare the STS performance of in children with CP and typical developing children. CP patients have difficulty in daily life activities due to muscle weakness, lack of muscle coordination, balance and postural control disorders. STS activity, which is one of the most frequently used activities in daily life, is a biomechanical activity in children with CP, requiring neuromuscular coordination and postural control outside of muscle strength. It is not enough to evaluate the muscle strength to evaluate the STS movement which is very important for these group, it is necessary to evaluate the balance of this movement of children with CP and the isolated muscle strengths (selective motor controls) of the lower extremity that we believe may affect this movement. There is not enough information about whether there is a relationship between the trunk controls and the selective motor controls of the lower extremities during the STS movement in children with CP. The information in the literature is limited to the fact that trunk control and muscle strength affect the balance during the STS movement. However, there is no study examining the relationship between selective motor control and trunk control during STS movement in children with CP.

This study, which includes selective motor control and trunk control, aims to eliminate this deficiency in the literature. In addition, the performance of the participants STS movement will be evaluated objectively with the test of the computerized balance device planned to be applied. In this study, to in children with CP; "Modified Ashworth Scale" to evaluate spasticity in the hip, knee and ankle, "Gross Motor Function Classification System" to determine gross motor levels, "Trunk Control Measurement Scale" to measure dynamic and static balance, "Gross Motor Function Measure-88's sitting sub-test" to assess seating function", "Selective Control Assesment of Lower Extremity" to assess the selective motor control of the knee and ankle muscles, the sit to stand test of the computerized postural analysis device will be applied to assess the duration of the STS movement and the deviations during the movement. The application time of the tests varies between 5-30 minutes.

For typical developing children, all tests except the Modified Ashworth Scale and the Gross Motor Function Classification System will be applied from tests applied to children with CP.

This study will evaluate the independence of children with CP in daily life activities and contribute to the correct planning of rehabilitation goals.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of spastic hemiplegic or diplegic cerebral palsy
2. Age between 4 - 10
3. Were having a level of 1 or 2 of GMFCS
4. Able to stand without any orthosis or special equipment
5. No orthopedic surgery or not having Botulinum Toxin-A injection in the last 6 months
6. Volunteer to study

Exclusion Criteria:

1. Having cognitive disorder
2. Uncontrolled epilepsy
3. Lower extremity contracture that may affect assessments

Ages: 4 Years to 10 Years | Sex: All
Age Groups: Child
Study Population: 16 spastic hemiplegic cerebral palsy patients, 12 spastic diplegic cerebral palsy patients between 4 - 10 years of age, and 32 healthy volunteer peers
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2020-01-04 (Estimated); Primary Completion 2020-03-04 (Estimated); Study Completion 2020-03-15 (Estimated)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | Baseline
  TCMS measures the state of balance on the support surface and the ability to actively move body parts during functional activities, which are the two components of trunk control. TCMS consists of 15 items in total that are scored on 2, 3 or 4 point ordinal scale and administered bilaterally in case of clinical relevance. The total TCMS score ranges from 0 to 58. A high score on this scale represents a better performance.

SECONDARY OUTCOMES:
Selective Control Assessment of the Lower Extremity | Baseline
  SCALE examines selective voluntary motor control in children with spastic CP. The SCALE tool assesses hip, knee, ankle, subtalar, and toe joints bilaterally.The SCALE tool assigns each joint a score from 0 to 2 points: 2 points, normal; 1 point, impaired; and 0 points, unable. The SCALE score is the sum of scoresfor each joint and assumes a 10 point maximum per limb.
Weight Transfer Time (sec) parameter of sit to stand test of Neurocome Balance Master | Baseline
  Evaluations will be done by Balance Master® device. The weight transfer time was defined as the length of time between the prompt to move and the moment when the COG shifted to over the feet.
Rising Index (%) parameter of sit to stand test of Neurocome Balance Master | Baseline
  The rising index, or the amount of force exerted by the legs to decelerate forward motion of the upper body during the rising phase, expressed as a percent of body weight.
Sway Velocity (deg/sec) | Baseline
  Center of gravity (COG) sway velocity, or the mean velocity of COG sway during the rise to stand and the first five seconds during standing, expressed in degree per second.
Sitting domain of Gross Motor Function Measurement-88 (GMFM-88) | Baseline
  Gross Motor Function Measurement evaluates motor functions in children with Cerebral Palsy. There is 88 items under 5 subdimensions (lying and rolling, sitting, crawling and kneeling, standing, walking-running-jumping. GMFM has a 4-point scoring system for each item. The higher the child gets, the more successful the child is in gross motor function

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag Saygi, Prof, Study Chair — Marmara University
Locations (1):
- Marmara University School of Medicine, Pendik Research and Education Hospital, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the principal investigator (DG). The data are not publicly available due to their containing information that could compromise the privacy of research participants.

REFERENCES:
- [Result] Fowler EG, Staudt LA, Greenberg MB, Oppenheim WL. Selective Control Assessment of the Lower Extremity (SCALE): development, validation, and interrater reliability of a clinical tool for patients with cerebral palsy. Dev Med Child Neurol. 2009 Aug;51(8):607-14. doi: 10.1111/j.1469-8749.2008.03186.x. Epub 2009 Feb 12. PMID 19220390
- [Result] Heyrman L, Molenaers G, Desloovere K, Verheyden G, De Cat J, Monbaliu E, Feys H. A clinical tool to measure trunk control in children with cerebral palsy: the Trunk Control Measurement Scale. Res Dev Disabil. 2011 Nov-Dec;32(6):2624-35. doi: 10.1016/j.ridd.2011.06.012. Epub 2011 Jul 14. PMID 21757321